CLINICAL TRIAL: NCT05813184
Title: Effect of Prenatal Antibiotics on Breast Milk Immune Function and on the Development of Neonatal Intestinal Immune System: the Role of IgA
Brief Title: Prenatal Antibiotics and Breast Milk / Neonatal IgA
Acronym: PAIGAN 1
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: Humanitas Hospital, Italy (Other)
Responsible Party: Principal Investigator, Carlo Pietrasanta, Senior Researcher, Principal Investigator, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Other Study IDs: 6530
Record Dates: First submitted 2023-04-02; First posted 2023-04-14 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Prenatal Exposure Delayed Effects; Antibiotic Prophylaxis; Dysbiosis; Neonatal Infection; Breast Milk; Noxious Influence, Affecting Fetus
Keywords: IgA; Prenatal antibiotics; breast milk; feces; neonatal immune system
MeSH Terms: conditions — Prenatal Exposure Delayed Effects; Dysbiosis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — fecal and breast milk microbiota
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Women not exposed to antibiotics throughout the entire duration of pregnancy
- Prenatal antibiotics: Women exposed to antibiotics for at least 7 days from the 32nd week of gestation
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Any antibiotic therapy administered > 7 days
  Groups: Prenatal antibiotics

SUMMARY:
In this biological study, the investigators will evaluate the levels of breast milk IgA, neonatal fecal IgA, and the composition of breast milk and fecal microbiota throughout the first 12 months of life in neonates born to mothers treated or not treated with prenatal antibiotics for at least 7 days after the 32nd weeks of gestation

DETAILED DESCRIPTION:
In a human cohort of women and their neonates, the investigators aim to evaluate the absolute amount of IgA in maternal breast milk and in neonatal feces in the presence (N=41 mother/infant pairs) or in the absence (N=41 mother/infant pairs) of exposure to prenatal ABX during the last period of pregnancy. Moreover, the investigators aim to evaluate, both in maternal breast milk and in neonatal feces, the composition of microbiota, and the proportion and composition of the IgA-coated and not-IgA- coated fractions of microbiota, by means of fluorescence-activated cell sorting (FACS) coupled with 16S rRNA sequencing of bacteria. Finally, the investigators will measure the concentration of the chemokine CCL28 on maternal serum and breast milk, as a soluble marker of activity of the entero-mammary pathway that is known to drive the migration of IgA producing plasma- cells from maternal mesenteric lymph nodes to the mammary gland.

All the analysis will be performed in mother-infant dyads with exclusive breastfeeding. Breast milk/serum/feces collection and analysis will be repeated at the following timepoints:

1. during the first week of neonatal life
2. at 1 month of life
3. at 3 months of life
4. at 8-12 months of life (or at the time of breastfeeding interruption), after the introduction of solid food in the infant's diet.

ELIGIBILITY:
Inclusion Criteria:

* expression of written informed consent
* an antibiotic treatment (any molecule) for at least 7 days consecutively after the 32 weeks of pregnancy (or the absence of exposure to any systemic antibiotic treatment during pregnancy for the control group)
* the intention to breastfeed their neonates as long as possible during the first year of life

Exclusion Criteria:

* absence of written informed consent
* the intention to formula feed exclusively (or the presence of significant maternal concerns about breastfeeding)
* a maternal antibiotic treatment shorter than 7 days
* the presence of pre-existing maternal immune-mediated disorders (including immunodeficiencies and chronic infectious diseases)
* a delivery at a gestational age < 34 weeks
* the administration of antibiotics to neonates after birth, within the first week of life.

Ages: 18 Years to 40 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnancy is a required condition
Study Population: pregnant women exposed or not exposed to antibiotics in the last trimester of pregnancy
Sampling Method: Non-Probability Sample
Enrollment: 82 (Estimated)
Dates: Start 2023-10-08 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-10-30 (Estimated)

PRIMARY OUTCOMES:
breast milk IgA | until 12 months of neonatal life
  concentration of IgA in breast milk

SECONDARY OUTCOMES:
fecal IgA | until 12 months of neonatal life
  concentration of IgA in neonatal feces
breast milk microbiota | until 12 months of neonatal life
  Composition of microbiota in breast milk and analysis of fractions coated or uncoated by IgA
fecal microbiota | until 12 months of neonatal life
  Composition of microbiota in breast milk and analysis of fractions coated or uncoated by IgA
maternal CCL28 | until 12 months of neonatal life
  concentration of CCL28 in maternal serum and breast milk

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Pietrasanta, MD,PhD, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided